CLINICAL TRIAL: NCT00950352
Title: Citicoline Treatment of Methamphetamine Dependence
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Perry Renshaw (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Perry Renshaw, Professor of Psychiatry, University of Utah
Organization: University of Utah (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 32808; CDP-1212
Record Dates: First submitted 2009-07-29; First posted 2009-07-31 (Estimated); Results first posted 2015-02-11 (Estimated); Last update posted 2015-02-11 (Estimated); Status verified 2015-02

CONDITIONS: Methamphetamine Dependence
Keywords: methamphetamine; Citicoline; CDP-Choline; Neuroimaging; MRI; Brain; MRS; DTI
MeSH Terms: interventions — Cytidine Diphosphate Choline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Citicoline (Experimental): In a double-blind randomization design, subjects with methamphetamine dependence will be treated with citicoline or placebo for 8-9 weeks.
  Interventions: Drug: Citicoline
- Placebo (Placebo Comparator): In a double-blind randomization design, subjects with methamphetamine dependence will be treated with citicoline or placebo for 8-9 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Citicoline — Subjects will be given 1g citicoline twice daily for a total of 8-9 weeks.
  Other Names: CDP-Choline
  Arms: Citicoline
Drug: Placebo — Subjects will be given 1 capsule of placebo twice daily for 8-9 weeks. They will be taking the same quantity as the citicoline group.
  Arms: Placebo

SUMMARY:
The purpose of the study is to determine if citicoline (a nutritional supplement) is effective in helping people reduce their dependence on methamphetamine. The investigators will use neuroimaging to look at the structure and chemical make up of the brain at the start of the study and after 8-9 weeks of treatment of citicoline or placebo.

DETAILED DESCRIPTION:
This is a prospective, randomized, double-blind, placebo-controlled study, in which we will systematically evaluate the therapeutic effects of citicoline, which may both increase dopamine and normalize cognitive and structural deficits in the brains of methamphetamine dependent subjects. Methamphetamine dependent subjects will undergo baseline and repeat cognitive assessments after 8-9 weeks of placebo or oral citicoline as a nutritional supplement. We will also evaluate the chemical and structural changes in brain regions identified by magnetic resonance spectroscopy (MRS), diffusion tension imaging (DTI) and cortical thickness, which in turn are expected to recover after 8-9 weeks of citicoline treatment. Specific brain regions of interest include the prefrontal cortices, temporal cortex, and the caudate/putamen all of which are known to be involved in the pathophysiology of methamphetamine dependence.

ELIGIBILITY:
Methamphetamine Dependent Subject Eligibility:

Inclusion Criteria:

* Subjects who use methamphetamine as their preferred drug of abuse.
* Subjects must be between the ages of 18 and 45 years.
* Subjects must have recent methamphetamine use (within 6 months of screening).
* Subjects must have an established residence and phone.
* Subjects must be able to give informed consent.

Exclusion Criteria:

* Significant current or past medical, neurological, or psychiatric co-morbidity including cardiovascular, renal, and endocrine disorder, as identified by medical history.
* Pregnant subjects - due to the unknown effects of MRI on a fetus. In addition, women of childbearing potential who will not practice a medically accepted method of contraception will be excluded. Female subjects who are of child-bearing potential will have to pass a urine pregnancy test before each visit.
* Subjects who, in the investigator's judgment, pose a current serious homicidal or suicidal risk.
* Subjects who will not likely be able to comply with the study protocol.
* Subjects who have any contraindication to an MR scan.
* Hypersensitivity to any of the study drugs or excipients
* Subjects with current DSM-IV diagnosis of a major mental illness. Major illness will be defined as Major Depression, Manic Depression, Schizophrenia, Dissociative Disorder, other psychotic illnesses, Attention-Deficit Hyperactivity Disorder, Post Traumatic Stress Disorder, Borderline Personality Disorder, Reactive Attachment Disorder, and Panic Disorder.
* Predominant alcohol or other substance dependence as preferred drug of abuse.
* Positive HIV test result.
* An individual having any pending legal or criminal charge or action, or who has pending or a reasonable potential for court involvement, or a person who is incarcerated or is in detention, or who is pending or having completed a competency evaluation or commitment procedure.

Healthy Control Subject Eligibility:

Inclusion Criteria:

* Subjects must be between the ages of 18 and 45 years.
* Subjects must be able to give informed consent.
* To have an established residence and phone.

Exclusion Criteria:

* Significant medical, neurological, or psychiatric disorders
* Pregnant subjects - due to the unknown effects of MRI on a fetus. In addition, women of childbearing potential who will not practice a medically accepted method of contraception will be excluded. Female subjects who are of child-bearing potential will have to pass a urine pregnancy test before each visit.
* Subjects who have any contraindication to an MR scan.
* Subjects unable to comply with protocol.
* Positive HIV test result.
* Positive urine drug screen.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 104 (Actual)
Dates: Start 2010-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Perry F Renshaw, MD, PhD, MBA, Principal Investigator — University of Utah
Locations (1):
- The Brain Institute of the University of Utah, Salt Lake City, Utah, United States

REFERENCES:
- See also: The Brain Institute — http://brain.utah.edu/
- See also: NIDA — http://www.nida.nih.gov/

RESULTS

PARTICIPANT FLOW:
Groups:
- Citicoline: 74 subjects with methamphetamine dependence were treated with citicoline for 8-9 weeks.
  Citicoline: Subjects were given 1g citicoline twice daily for a total of 8-9 weeks.
- Placebo: 32 subjects with methamphetamine dependence were treated with placebo for 8-9 weeks.
  Placebo: Subjects were given 1 g of placebo twice daily for 8-9 weeks. They will be taking the same quantity as the citicoline group.
Period: Overall Study
Arm/Group | Citicoline | Placebo
Started | 72 | 32
Completed | 30 | 21
Not Completed | 42 | 11

BASELINE CHARACTERISTICS:
Groups:
- Placebo: 32 subjects with methamphetamine dependence were treated with citicoline for 8-9 weeks.
  Placebo: Subjects were given 1 capsule of placebo twice daily for 8-9 weeks. They will be taking the same quantity as the citicoline group.
- Total: Total of all reporting groups
Arm/Group | Citicoline | Placebo | Total
Number analyzed (Participants) | 72 | 32 | 104
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 72 | 32 | 104
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.9 (6.8) | 31.4 (7.1) | 32.4 (6.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 14 | 47
  Male | 39 | 18 | 57
Region of Enrollment [Number; unit: participants]
  United States | 72 | 32 | 104

OUTCOME MEASURES:

1. Primary Outcome: Methamphetamine Dependent Subjects Treated With Citicoline vs Placebo
Description: Total Amount of Methamphetamine consumed by the participants after 8-9 weeks of treatment. Methamphetamine was assessed twice weekly.
Time Frame: 8 weeks, assessed twice weekly starting week1
Measure: Mean (Standard Deviation); unit: total amount consumed in grams
Groups:
- Placebo: Subjects will be given 1 g of placebo twice daily for 8-9 weeks. They will be taking the same quantity as the citicoline group.
Arm/Group | Citicoline | Placebo
Number analyzed (Participants) | 30 | 21
total amount consumed in grams | 0.3025 (0.16498) | 0.3850 (0.34547)

2. Secondary Outcome: Testing if Citicoline Administration Will be Associated With Significant Improvements in Neuropsychological Performance.
Description: Cognitive measurement tests will be employed.
Time Frame: Neuropsychological testing will occur at week 0 and week 8/9
Reporting Status: Not Posted

3. Secondary Outcome: Testing if Neuroimaging Measures Will Show Significant Improvements in Brain Chemical and Structural Parameters After 8-9 Weeks of Citicoline Treatment in Methamphetamine Dependent Subjects.
Description: Phosphorus-31 ((31)P) magnetic resonance spectroscopy (MRS) was used to evaluate changes in mitochondrial high energy phosphates, including phosphocreatine (PCr) and β-nucleoside triphosphate (β-NTP, primarily ATP in brain) levels.
Time Frame: Neuroimaging will occur at week 0 and week 8/9
Reporting Status: Not Posted

4. Secondary Outcome: Testing if Improvements in Cognitive Function as Well as Brain Chemical and Structural Parameters Will be Associated With Greater Reductions in Drug Use.
Description: Self report drug use and mood will be evaluated at each study visit throughout the course of the study. Also, urine samples will be collected twice a week for drugs of abuse testing.
Time Frame: Throughout the course of the study
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Citicoline | Placebo
Serious Adverse Events (participants affected / at risk) | 2/72 | 0/32
Other Adverse Events (participants affected / at risk) | 10/72 | 14/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Citicoline (N=72) | Placebo (N=32)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0) — A 36 year old male study participant had a suicide attempt during the eight week of the study. He ingested five Atenolol tablets (100g). Serious adverse event was unexpected and not related to the study medication (citicholine or placebo).
Sepsis (Infections and infestations) | 1 (1) | 0 (0) — Subject was hospitalized for sepsis due to an untreated UTI. The serious adverse event was unexpected and not related to the study medication (citicholine or placebo)
OTHER ADVERSE EVENTS (reported when occurring in more than 2.7% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Citicoline (N=72) | Placebo (N=32)
Gatsrointestinal symptoms (Gastrointestinal disorders) | 2 (2) | 4 (4)
General (Weight loss, Headache, Cold/flu-lie symptoms, fatigue, pulmonary) (General disorders) | 6 (6) | 6 (6) — Symptoms were assessed as "General" irrespective of the actual event
Psychiatric (Psychiatric disorders) | 2 (2) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No